CLINICAL TRIAL: NCT05322408
Title: A Phase I Study of HCW9218, a Bifunctional TGF-B; Antagonist/IL-15 Protein Complex, in Select Advanced Solid Tumors After Failing at Least Two Prior Therapies
Brief Title: HCW9218 in Select Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS143
Record Dates: First submitted 2022-03-31; First posted 2022-04-11 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administer HCW9218 (Experimental): Administer HCW9218 as monotherapy at assigned dose by SC injection once every 3 weeks. Dose Level
  -1 - 0.1 mg/kg
  1. - (start) 0.25 mg/kg
  2. - 0.5 mg/kg
  3. - 0.8 mg/kg
  4. - 1.2 mg/kg
  Interventions: Drug: HCW9218

INTERVENTIONS:
Drug: HCW9218 — HCW9218 at the assigned dose level is administered as a subcutaneous injection once every 3 weeks for a minimum of 2 treatment cycles unless medically contraindicated.
  Other Names: Monotherapy

SUMMARY:
This is a single center, Phase I dose finding study of HCW9218 for the treatment of advanced/metastatic solid tumor cancer (except pancreatic and primary brain cancers). HCW9218 is a novel bi-functional fusion protein complex administered by subcutaneous (SC) injection. It is comprised of a soluble fusion of two human TGFβRII domains, human tissue factor, and human IL-15, and a second soluble fusion of two human TGFβRII domains and a sushi domain of human IL-15Rα. HCW9218 activates IL-15R signaling on effector immune cells and the dimeric TGFβRII functions as a "trap" for all three human TGF-β isoforms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced/metastatic solid tumor cancer (except pancreatic and primary brain cancers), has failed at least 2 prior lines of therapy given either in the recurrent or metastatic setting and must be refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.
* Measurable disease per RECIST v 1.1.
* Acute effects of any prior therapy must have resolved to baseline or Grade ≤1 NCI CTCAE v5 except for AEs not constituting a safety risk by enrolling Investigator judgment.
* Age 18 years or older at the time of consent.
* ECOG Performance Status 0 or 1.
* Evidence of adequate organ function within 14 days prior to enrollment as defined in Section 4.1.6.
* Adequate pulmonary function with PFTs >50% FEV1 if symptomatic or known impairment.
* Sexually active persons of child-bearing potential or with partners of childbearing potential must agree to use a highly effective form of contraception (refer to Section 4.1.10 for acceptable methods) for at least 28 days after the last dose of HCW9218.
* Provides voluntary written consent prior to the performance of any research related activity.

Exclusion Criteria:

* Pregnant or breastfeeding.
* History of clinically significant vascular disease, including any of the following within 6 months prior to start of study treatment: MI or unstable angina, percutaneous coronary intervention, bypass grafting, ventricular arrhythmia requiring medication, stroke or transient ischemic attack, symptomatic peripheral arterial disease.
* Marked baseline prolongation of QT/QTc interval (e.g., demonstration of a QTc interval greater or equal to 470 milliseconds by Fridericia's correction).
* Known or suspected untreated CNS metastases.
* Anti-cancer treatment including surgery, radiotherapy, chemotherapy, other immunotherapy, or investigational therapy within 14 days before treatment start.
* Other prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the subject is currently in complete remission, or any other cancer from which the subject has been disease-free for 3 years after surgical treatment.
* Known hypersensitivity or history of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study.
* Prior therapy with TGF-β antagonist, IL-15 or analogs.
* Concurrent use of St. John's wort and and/or other herbal CYP modulators within 7 days of Day 1. Must agree to not use during study treatment through the end of treatment visit to be eligible.
* Known autoimmune disease requiring active treatment. Persons with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
* Prior organ allograft or allogeneic transplantation.
* Known HIV-positive or AIDS.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Other illness or a medical issue that in the opinion of the Investigator would exclude the subject from participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota
Locations (1):
- Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HCW9218 Dose Level -1; HCW9218 Dose Level 1; HCW9218 Dose Level 2; HCW9218 Dose Level 3; HCW9218 Dose Level 4: Administer HCW9218 as monotherapy at assigned dose by SC injection once every 3 weeks.
  Dose Level
  -1 - 0.1 mg/kg
  1. - (start) 0.25 mg/kg
  2. - 0.5 mg/kg
  3. - 0.8 mg/kg
  4. - 1.2 mg/kg
  HCW9218: HCW9218 at the assigned dose level is administered as a subcutaneous injection once every 3 weeks for a minimum of 2 treatment cycles unless medically contraindicated.
Period: Overall Study
Arm/Group | HCW9218 Dose Level -1 | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Started | 0 | 3 | 3 | 3 | 9
Completed | 0 | 3 | 3 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 6 | 14
  >=65 years | 1 | 0 | 0 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 6 | 9
  Male | 2 | 2 | 2 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 2 | 3 | 3 | 7 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Dose Finding Component is to Determine the Maximum Tolerated Dose (MTD) of HCW9218
Description: Given that little to no toxicity is expected, the MTD will be determined using an adaptation of the continual reassessment method (CRM) (O'Quigley, 1996) starting with 1 patient cohorts.
Time Frame: through study completion, an average of 12 months
Measure: Number; unit: mg/kg
Groups:
- Administer HCW9218: Administer HCW9218 as monotherapy at assigned dose by SC injection once every 3 weeks. Dose Level
  -1 - 0.1 mg/kg
  1. - (start) 0.25 mg/kg
  2. - 0.5 mg/kg
  3. - 0.8 mg/kg
  4. - 1.2 mg/kg
  HCW9218: HCW9218 at the assigned dose level is administered as a subcutaneous injection once every 3 weeks for a minimum of 2 treatment cycles unless medically contraindicated.
Arm/Group | Administer HCW9218
Number analyzed (Participants) | 18
mg/kg | 1.2

2. Secondary Outcome: Estimate Response Rate (Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Response rate will be estimated by a simple proportion with 95% confidence limits if sufficient numbers exist
Time Frame: 3 months after 1st dose
Measure: Count of Participants; unit: Participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 9
Participants | 1 | 1 | 1 | 5

3. Secondary Outcome: Estimate Response Rate (Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Response rate will be estimated by a simple proportion with 95% confidence limits if sufficient numbers exist
Time Frame: 6 months after 1st dose
Measure: Count of Participants; unit: Participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 1 | 2 | 2 | 6
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Estimate Response Rate (Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Response rate will be estimated by a simple proportion with 95% confidence limits if sufficient numbers exist
Time Frame: 12 months after 1st dose
Population: Unable to analyze participants in dose level 1 due to all cause mortality.
Measure: Count of Participants; unit: Participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 1 | 1 | 1 | 5
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Estimate Progression of Overall Survival (OS)
Description: Estimated with Kaplan-Meier curves
Time Frame: 6 months after 1st dose
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 9
Percentage of participants | 67 [5 to 95] | 67 [5 to 95] | 67 [5 to 95] | 78 [36 to 94]

6. Secondary Outcome: Estimate Progression Free Survival (PFS)
Description: Estimated with Kaplan-Meier curves
Time Frame: 6 months after 1st dose
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 9
Percentage of participants | 33 [1 to 77] | 0 [0 to 100] | 0 [0 to 100] | 11 [1 to 39]

7. Secondary Outcome: Estimate Progression Free Survival (PFS)
Description: Estimated with Kaplan-Meier curves
Time Frame: 1 year after 1st dose
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 9
Percentage of participants | 33 [1 to 77] | 0 [0 to 100] | 0 [0 to 100] | 11 [1 to 39]

8. Secondary Outcome: Estimate Progression of Overall Survival (OS)
Description: Estimated with Kaplan-Meier curves
Time Frame: 1 year after 1st dose
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 9
Percentage of participants | 33 [1 to 77] | 33 [1 to 77] | 33 [1 to 77] | 67 [28 to 88]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HCW9218 Dose Level 1 | HCW9218 Dose Level 2 | HCW9218 Dose Level 3 | HCW9218 Dose Level 4
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 6/9
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 0/3 | 4/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCW9218 Dose Level 1 (N=3) | HCW9218 Dose Level 2 (N=3) | HCW9218 Dose Level 3 (N=3) | HCW9218 Dose Level 4 (N=9)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Ascites (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Other, specify - C.Diff Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Obstruction (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic obstruction - Partial bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCW9218 Dose Level 1 (N=3) | HCW9218 Dose Level 2 (N=3) | HCW9218 Dose Level 3 (N=3) | HCW9218 Dose Level 4 (N=9)
Injection site reaction (General disorders) | 3 (11) | 3 (15) | 3 (17) | 9 (44)
Flu like symptoms (General disorders) | 1 (1) | 3 (7) | 3 (14) | 8 (22)
Fever (General disorders) | 1 (2) | 1 (1) | 2 (2) | 8 (13)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (8)
Disease progression (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (6) | 3 (6) | 3 (7) | 8 (19)
White blood cell decreased (Investigations) | 0 (0) | 1 (2) | 3 (5) | 5 (8)
Activated partial thromboplastin time prolonged (Investigations) | 2 (5) | 0 (0) | 1 (1) | 5 (16)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 6 (10)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 2 (2) | 5 (11)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (2) | 3 (7)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 5 (10)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
INR increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 2 (6)
Weight gain (Investigations) | 1 (4) | 0 (0) | 1 (1) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 1 (3) | 5 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0) | 2 (2) | 6 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (6) | 1 (1) | 2 (6) | 6 (13)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (2) | 4 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 3 (5) | 2 (6) | 5 (11)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (8)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (3) | 0 (0) | 3 (9)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (5)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (6)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT05322408/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05322408/ICF_001.pdf